CLINICAL TRIAL: NCT01494688
Title: Open-Label, Multicenter, Dose Escalation Phase Ia/Ib Study With Expansion Phase to Evaluate Safety, Pharmacokinetics and Activity of RO5509554, Administered as an Intravenous Infusion as Monotherapy and in Combination With Paclitaxel in Patients With Advanced Solid Tumors
Brief Title: A Study of RO5509554 as Monotherapy and in Combination With Paclitaxel in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP27772; 2011-003394-28 (EudraCT Number)
Record Dates: First submitted 2011-12-02; First posted 2011-12-19 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Paclitaxel; emactuzumab

ARMS (4):
- Part 1 - Dose Escalation: RO5509554 (Experimental): Participants will receive a single, low dose of 100 milligrams (mg) RO5509554 in 7-day PK run-in period (Cycle 0), followed by dose escalation from Day 1 of Cycle 1. RO5509554 will be escalated as monotherapy in approximately 6 cohorts with dose increments between cohorts of up to 100 percent (%). The doses will be escalated further until MTD/OBD as single agent is reached.
  Interventions: Drug: RO5509554
- Part 1 - Dose Escalation: RO5509554 + Paclitaxel (Experimental): RO5509554 will be administered in combination with a fixed dose of weekly (QW) paclitaxel (80 milligrams per square meter [mg/m^2]). The starting dose for RO5509554 in combination with paclitaxel will be 2 dose levels below to that of the highest dose of monotherapy RO5509554. Escalation of RO5509554 in combination with QW paclitaxel will start in a standard 3 + 3 design until MTD/OBD as combination dose is reached. If the initial combination is not tolerated, further cohorts will be dosed with the same dose of paclitaxel and lower dose of RO5509554. If insufficient safety, pharmacokinetic or pharmacodynamic data have been collected at the MTD/OBD, up to an additional 4 participants may be enrolled at that dose level.
  Interventions: Drug: Paclitaxel; Drug: RO5509554
- Part 2 - Expansion Cohort: RO5509554 (Experimental): Participants will receive RO5509554 1000 mg Q2W, Q3W or initial biweekly followed by monthly maintenance.
  Interventions: Drug: RO5509554
- Part 2 - Expansion Cohort: RO5509554 + Paclitaxel (Experimental): Participants will receive RO5509554 1000 mg Q2W in combination with a fixed dose of QW paclitaxel (80 mg/m^2).
  Interventions: Drug: Paclitaxel; Drug: RO5509554

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel, at a dose of 80 mg/m^2 will be administered QW for up to 12 weeks.
  Arms: Part 1 - Dose Escalation: RO5509554 + Paclitaxel; Part 2 - Expansion Cohort: RO5509554 + Paclitaxel
Drug: RO5509554 — RO5509554 will be administered Q2W, Q3W or initial biweekly followed by monthly maintenance as intravenous (IV) infusion until disease progression, unacceptable toxicity, death or participant refusal, whichever occurs first.
  Other Names: RG7155

SUMMARY:
This open-label, multicenter, dose-escalation study will assess the safety, tolerability, pharmacokinetics and pharmacodynamics of RO5509554 in participants with advanced solid tumors which are not amenable to standard treatment. In Part I (Dose Escalation), multiple ascending doses of RO5509554 will be administered as monotherapy in participants with solid tumors. Participants with locally advanced and/or metastatic ovarian (including fallopian tube) and breast carcinoma will receive multiple ascending doses of RO5509554 in combination with paclitaxel. In Part II (Expansion Cohort), RO5509554 will be administered as monotherapy to participants with locally advanced and/or metastatic Pigmented Villonodular Synovitis (PVNS)/Tenosynovial Giant Cell Tumor (TGCT), soft tissue sarcoma or malignant mesothelioma, ovarian (including fallopian tube), endometrial or breast cancer and pancreatic cancer. Participants with Human Epidermal Growth Factor Receptor 2 (HER2)/neu negative breast cancer will receive RO5509554 in combination with paclitaxel. Anticipated time on study treatment is until disease progression, unacceptable toxicity, death or participant refusal, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced and/or metastatic solid tumors which are not amenable to standard therapy, with exceptions as defined in exclusion criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Measurable disease according to RECIST criteria version 1.1
* Adequate bone marrow, cardiac, liver and renal function

Exclusion Criteria:

* Participants with histologically proven Hepatocellular Carcinoma (HC), Non Small Cell Lung Cancer (NSCLC), Small Cell Lung Cancer (SCLC), gastric cancer, malignant melanoma, nonmetastatic and locally controlled PVNS/TGCT
* Participants with known auto-immune disease
* Known or suspected central nervous system (CNS) metastases including leptomeningeal metastasis; participants with radiologically stable, asymptomatic previously irradiated lesion are eligible provided participant is greater than or equal to (>/=) 4 weeks beyond completing cranial irradiation and >/= 3 weeks of corticosteroid therapy
* Significant, uncontrolled concomitant diseases, including significant cardiovascular or pulmonary disease
* Prior chemotherapy, radiotherapy (other than short cycle of palliative radiotherapy for bone pain), any investigational agent or immunotherapy within 28 days of first receipt of study drug
* Prior corticosteroids as anti-cancer therapy within minimum of 14 days of first receipt of study drug
* Poorly controlled type 1 or type 2 diabetes mellitus
* Prior toxicities from chemotherapy or radiotherapy which have not regressed to Grade less than or equal to (</=) 1 severity National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 or later versions
* Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) infection
* Pulmonary embolism or any other thrombo-embolic event within 6 months prior to study entry
* History of hematological malignancy within the last 5 years prior to study entry
* Participant requires high dose corticosteroid treatment ( i.e. greater than (>) 20 mg dexamethasone a day or equivalent for > 7 consecutive days)
* Any surgical procedure, including the required baseline tumor biopsy, within less than 14 days of first receipt of study drug. Major surgery within 28 days of first receipt of study drug
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2011-12-20 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events | Baseline up to 28 days after last dose (approximately 48 months)
Part 1: Maximum Tolerated Dose (MTD)/Optimal Biological Dose (OBD) of RO5509554 as a Single Agent and in Combination With Paclitaxel | Cycle 1 Day 1 (cycle length = 14 or 21 days) up to 28 days

SECONDARY OUTCOMES:
Part 2: Change in Colony Stimulating Factor-1 (CSF-1) Serum Level For Every 2 Weeks (Q2W) Schedule | Pre-dose (0 hour [h]), 2, 5, 24, 72 or 96, 168, 216 and 264 h post-dose Cycles 1 & 4; 0 h & any time on Day 8 Cycle 2; 0 h Cycle 3; 0 h Cycle 5 & any time during 28 days follow-up; 0 h Cycle 6 onward up to 48 months [Each cycle=14 days]
Part 2: Change in CSF-1 Serum Level For Every 3 Weeks (Q3W) Schedule | Pre-dose (0 h), 3, 24, 72, 168, 264, 312, 432 & 480 h post-dose Cycles 1 & 4; 0 h Cycles 2 & 3; 0 h Cycle 5 & any time during 28 days follow-up; 0 h Cycle 6 onward up to 48 months [Each cycle=21 days]
Part 2: Change in CSF-1 Serum Level For Initial Q2W Followed by Monthly Maintenance Schedule | Pre-dose (0 h), 2, 5, 24, 72 or 96, 168, 216 & 264 h post-dose Cycle 1; 0 h & any time on Day 8 Cycle 2; 0 h & 5, 24, 72 or 96, 168, 264, 336, 432, 504 & 576 h post-dose Cycle 3; 0 h Cycle 4 onward up to 48 months [Each cycle=14 or 30 days]
Change in Circulating Monocytes Subset in Whole Blood For Q2W Schedule | 0,2,5,24,72 or 96,168,216 & 264 h post-dose Cycle 1; 0 h Day 1, any time Day 8 Cycle 2; 0 h Cycles 3 & 5; 0,5,72 or 96,168,216 & 264 h post-dose Cycle 4 & any time during 28 days follow-up; 0 h Cycle 6 onward up to 48 months [Each cycle=14 days]
Change in Circulating Monocytes Subset in Whole Blood For Q3W Schedule | 0, 3, 24, 72, 168, 264, 312, 432 & 480 h post-dose Cycle 1; 0 h Cycles 2 & 3; 0, 3, 72, 168, 264, 312, 432 & 480 h post-dose Cycle 4; 0 h Cycle 5 & any time during 28 days follow-up; 0 h Cycle 6 onward up to 48 months [Each cycle=21 days]
Change in Circulating Monocytes Subset in Whole Blood For Initial Q2W Followed by Monthly Maintenance Schedule | Pre-dose (0 h), 2, 5, 24, 72 or 96, 168, 216 & 264 h post-dose Cycle 1; 0 h & any time on Day 8 Cycle 2; 0h & 5, 24, 72 or 96, 168, 264, 336, 432, 504 & 576 h post-dose Cycle 3; 0 h Cycle 4 onward up to 48 months [Each cycle=14 or 30 days]
Pharmacokinetics of RO5509554: Area Under the Plasma concentration-Time Curve (AUC) for Q2W Schedule | Pre-dose(0 h),end of infusion(EOI)(over 1.5 h)& 3,4,5,6,24,72 or 96,168,216&264 h post-dose Cycle 1;0 h & EOI Cycles 2,3&5; 0 h,EOI &2,3,4,5,6,24,72 or 96,168,216&264 h post-dose at Cycle 4;0 h,EOI Cycle 6 onward up to 48 months [Each cycle=14 days]
Pharmacokinetics of RO5509554: AUC for Q3W Schedule | Pre-dose (0 h), EOI (over 1.5 h) and 3, 24, 72, 168, 264, 312, 432 and 480 h post-dose Cycles 1 and 4; pre-dose (0 h) and EOI Cycles 2, 3 and 5; pre-dose (0 h), EOI Cycle 6 onwards up to 48 months [Each cycle=21 days]
Pharmacokinetics of RO5509554: AUC for Initial Q2W Followed by Monthly Maintenance Schedule | Pre-dose(0 h),EOI(over 1.5 h), 3, 5, 24, 72 or 96, 168, 216, 264 h post-dose Cycle 1; 0 h & EOI Cycle 2; 0 h, EOI & 3, 5, 24, 72 or 96, 168, 264, 336, 432, 504, 576 h post-dose Cycle 3; 0 h & EOI Cycle 4 onward up to 48 months [Each cycle=14 or 30 days]
Pharmacokinetics of RO5509554: Maximum Observed Plasma concentration (Cmax) for Q2W Schedule | Pre-dose(0 h), EOI (over 1.5 h) & 3,4,5,6,24,72 or 96,168,216&264 h post-dose Cycle 1;0 h & EOI Cycles 2,3&5; 0 h,EOI &2,3,4,5,6,24,72 or 96,168,216&264 h post-dose at Cycle 4;0 h,EOI Cycle 6 onward up to 48 months [Each cycle=14 days]
Pharmacokinetics of RO5509554: Cmax for Q3W Schedule | Pre-dose (0 h), EOI (over 1.5 h) and 3, 24, 72, 168, 264, 312, 432 and 480 h post-dose Cycles 1 and 4; pre-dose (0 h) and EOI Cycles 2, 3 and 5; pre-dose (0 h), EOI Cycle 6 onwards up to 48 months [Each cycle=21 days]
Pharmacokinetics of RO5509554: Cmax for Initial Q2W Followed by Monthly Maintenance Schedule | Pre-dose(0 h),EOI(over 1.5 h), 3, 5, 24, 72 or 96, 168, 216, 264 h post-dose Cycle 1; 0 h & EOI Cycle 2; 0 h, EOI & 3, 5, 24, 72 or 96, 168, 264, 336, 432, 504, 576 h post-dose Cycle 3; 0 h & EOI Cycle 4 onward up to 48 months [Each cycle=14 or 30 days]
Pharmacokinetics of RO5509554: Half-life (t1/2) for Q2W Schedule | Pre-dose(0 h), EOI (over 1.5 h) & 3,4,5,6,24,72 or 96,168,216&264 h post-dose Cycle 1;0 h & EOI Cycles 2,3&5; 0 h,EOI &2,3,4,5,6,24,72 or 96,168,216&264 h post-dose at Cycle 4;0 h,EOI Cycle 6 onward up to 48 months [Each cycle=14 days]
Pharmacokinetics of RO5509554: t1/2 for Q3W Schedule | Pre-dose (0 h), EOI (over 1.5 h) and 3, 24, 72, 168, 264, 312, 432 and 480 h post-dose Cycles 1 and 4; pre-dose (0 h) and EOI Cycles 2, 3 and 5; pre-dose (0 h), EOI Cycle 6 onwards up to 48 months [Each cycle=21 days]
Pharmacokinetics of RO5509554: t1/2 Initial Q2W Followed by Monthly Maintenance Schedule | Pre-dose(0 h),EOI(over 1.5 h), 3, 5, 24, 72 or 96, 168, 216, 264 h post-dose Cycle 1; 0 h & EOI Cycle 2; 0 h, EOI & 3, 5, 24, 72 or 96, 168, 264, 336, 432, 504, 576 h post-dose Cycle 3; 0 h & EOI Cycle 4 onward up to 48 months [Each cycle=14 or 30 days]
Pharmacokinetics of RO5509554: Systemic Clearance (CL) for Q2W Schedule | Pre-dose(0 h), EOI (over 1.5 h) & 3,4,5,6,24,72 or 96,168,216&264 h post-dose Cycle 1;0 h & EOI Cycles 2,3&5; 0 h,EOI &2,3,4,5,6,24,72 or 96,168,216&264 h post-dose at Cycle 4;0 h,EOI Cycle 6 onward up to 48 months [Each cycle=14 days]
Pharmacokinetics of RO5509554: CL for Q3W Schedule | Pre-dose (0 h), EOI (over 1.5 h) and 3, 24, 72, 168, 264, 312, 432 and 480 h post-dose Cycles 1 and 4; pre-dose (0 h) and EOI Cycles 2, 3 and 5; pre-dose (0 h), EOI Cycle 6 onwards up to 48 months [Each cycle=21 days]
Pharmacokinetics of RO5509554: CL for Initial Q2W Followed by Monthly Maintenance Schedule | Pre-dose(0 h),EOI(over 1.5 h), 3, 5, 24, 72 or 96, 168, 216, 264 h post-dose Cycle 1; 0 h & EOI Cycle 2; 0 h, EOI & 3, 5, 24, 72 or 96, 168, 264, 336, 432, 504, 576 h post-dose Cycle 3; 0 h & EOI Cycle 4 onward up to 48 months [Each cycle=14 or 30 days]
Change in Pharmacodynamic Markers: Dermal Macrophages Expressing CD68/CD163 and Colony Stimulating Factor-1 Receptor (CSF-1R) in Paired Skin Biopsies | Baseline, Day 1 Cycle 2 pre-dose (0 h), Day 8 Cycle 2 [Each Cycle = 14 or 21 days]
Change in Pharmacodynamic Markers: Dermal Macrophages Expressing CD68/CD163 and CSF-1R in Paired Tumor Biopsies | Day -21 to -14, pre-dose (0 h) Day 1 Cycle 3 [Each Cycle = 14 or 21 days]
Change in Pharmacodynamic Markers: Tumor associated Macrophages (TAM) expressing Cells in Surrogate/Tumor Tissue (in Paired Tumor Biopsies) | Day -21 to -14, pre-dose (0 h) Day 1 Cycle 3 [Each Cycle = 14 or 21 days]
Standard Uptake Value of 18F Fluoro-Deoxy-Glucose (FDG), as Assessed Using Positron Emission Tomography (PET) Imaging | Baseline up to Cycle 3 Days 1 or 7 (Cycle length = 14 or 21 days)
Part 1: Recommended Phase II Dose (RP2D) of RO5509554 | Cycle 1 Day 1 (cycle length = 14 or 21 days) up to 28 days
Percentage of Participants With Objective Response (OR) Assessed According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | From screening to disease progression, death, withdrawal, or end of study; assessed at screening (within 3 weeks before first dose of study drug) then Day 1 of every third cycle (Each Cycle=14 or 21 days) until end of treatment (approximately 48 months)
Percentage of Participants With Clinical Benefit Assessed According to RECIST Version 1.1 | From screening to disease progression, death, withdrawal, or end of study; assessed at screening (within 3 weeks before first dose of study drug) then Day 1 of every third cycle (Each Cycle=14 or 21 days) until end of treatment (approximately 48 months)
Progression Free Survival (PFS) Assessed According to RECIST Version 1.1 | From screening to disease progression, death, withdrawal, or end of study; assessed at screening (within 3 weeks before first dose of study drug) then Day 1 of every third cycle (Each Cycle=14 or 21 days) until end of treatment (approximately 48 months)
Duration of Response Assessed According to RECIST Version 1.1 | From screening to disease progression, death, withdrawal, or end of study; assessed at screening (within 3 weeks before first dose of study drug) then Day 1 of every third cycle (Each Cycle=14 or 21 days)) until end of treatment (approximately 48 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Univ of Pennsylvania Med Ctr, Philadelphia, Pennsylvania
- France (5):
  - Institut Bergonie; Oncologie, Bordeaux
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Institut Curie; Oncologie Medicale, Paris
  - Ico Rene Gauducheau; Oncologie, Saint-Herblain
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse

REFERENCES:
- [Derived] Cassier PA, Italiano A, Gomez-Roca C, Le Tourneau C, Toulmonde M, D'Angelo SP, Weber K, Loirat D, Jacob W, Jegg AM, Michielin F, Christen R, Watson C, Cannarile M, Klaman I, Abiraj K, Ries CH, Weisser M, Ruttinger D, Blay JY, Delord JP. Long-term clinical activity, safety and patient-reported quality of life for emactuzumab-treated patients with diffuse-type tenosynovial giant-cell tumour. Eur J Cancer. 2020 Dec;141:162-170. doi: 10.1016/j.ejca.2020.09.038. Epub 2020 Nov 5. PMID 33161240
- [Derived] Gomez-Roca CA, Italiano A, Le Tourneau C, Cassier PA, Toulmonde M, D'Angelo SP, Campone M, Weber KL, Loirat D, Cannarile MA, Jegg AM, Ries C, Christen R, Meneses-Lorente G, Jacob W, Klaman I, Ooi CH, Watson C, Wonde K, Reis B, Michielin F, Ruttinger D, Delord JP, Blay JY. Phase I study of emactuzumab single agent or in combination with paclitaxel in patients with advanced/metastatic solid tumors reveals depletion of immunosuppressive M2-like macrophages. Ann Oncol. 2019 Aug 1;30(8):1381-1392. doi: 10.1093/annonc/mdz163. PMID 31114846
- [Derived] Cassier PA, Italiano A, Gomez-Roca CA, Le Tourneau C, Toulmonde M, Cannarile MA, Ries C, Brillouet A, Muller C, Jegg AM, Broske AM, Dembowski M, Bray-French K, Freilinger C, Meneses-Lorente G, Baehner M, Harding R, Ratnayake J, Abiraj K, Gass N, Noh K, Christen RD, Ukarma L, Bompas E, Delord JP, Blay JY, Ruttinger D. CSF1R inhibition with emactuzumab in locally advanced diffuse-type tenosynovial giant cell tumours of the soft tissue: a dose-escalation and dose-expansion phase 1 study. Lancet Oncol. 2015 Aug;16(8):949-56. doi: 10.1016/S1470-2045(15)00132-1. Epub 2015 Jul 12. PMID 26179200
- [Derived] Ries CH, Cannarile MA, Hoves S, Benz J, Wartha K, Runza V, Rey-Giraud F, Pradel LP, Feuerhake F, Klaman I, Jones T, Jucknischke U, Scheiblich S, Kaluza K, Gorr IH, Walz A, Abiraj K, Cassier PA, Sica A, Gomez-Roca C, de Visser KE, Italiano A, Le Tourneau C, Delord JP, Levitsky H, Blay JY, Ruttinger D. Targeting tumor-associated macrophages with anti-CSF-1R antibody reveals a strategy for cancer therapy. Cancer Cell. 2014 Jun 16;25(6):846-59. doi: 10.1016/j.ccr.2014.05.016. Epub 2014 Jun 2. PMID 24898549